CLINICAL TRIAL: NCT06965465
Title: A PHASE 1, RANDOMIZED, DOUBLE BLIND, SPONSOR-OPEN, PLACEBOCONTROLLED, SINGLE DOSE ESCALATION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SUBCUTANEOUS ADMINISTRATION OF PF-07999415 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Called PF-07999415 Are Tolerated and Act in the Body in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C5671001; 2024-520380-13-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PF-07999415 (Experimental)
  Interventions: Biological: PF-07999415
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: PF-07999415 — Participants will receive single doses of PF-07999415.
  Arms: PF-07999415
Drug: Placebo — Participants will receive matching placebo.
  Arms: Placebo

SUMMARY:
The purpose of this clinical study is to learn about the safety and effects of the study medicine (called PF-07999415) in healthy adult participants.

This study is seeking volunteers aged 18 to 65 years old who do not have any major health issues.

Some participants in this study will receive a single dose of PF-07999415 as a shot in the thigh, abdomen, or arm at the study clinic. Afterward, participants will stay in a hospital-like setting for 2 weeks, where they will be monitored for reactions to the study medicine.

The study team will compare the experiences of people receiving PF-07999415 to those of the people who do not. This will help the study team decide if PF-07999415 is safe.

Participants will take part in this study for 3 to 7 months. During this time, participants will stay at the healthcare facility for 2 weeks and then come back for study visits every 2 weeks until completing the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants of non-childbearing potential aged 18 to 65 years, inclusive, at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body Mass Index (BMI) of 18-33 kg/m2 and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, dermatological, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Previous administration of an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events. | First dose (Day 1) to up to final follow-up visit (Day 85)

SECONDARY OUTCOMES:
Area under the concentration-time profile from time 0 to the time of the last quantifiable concentration (AUClast) for PF-07999415 | First dose (Day 1) to up to final follow-up visit (Day 85)
Maximum observed concentration (Cmax) for PF-07999415 | First dose (Day 1) to up to final follow-up visit (Day 85)
Time to maximum observed concentration (Tmax) for PF-07999415 | First dose (Day 1) to up to final follow-up visit (Day 85)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5671001